CLINICAL TRIAL: NCT01849926
Title: Ibuprofen Versus Mecillinam for Uncomplicated Cystitis in Adult, Non-pregnant Women
Brief Title: Ibuprofen Versus Mecillinam for Uncomplicated Cystitis
Acronym: IMUTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: University of Bergen (Other); Lund University (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Lindbaek, Professor dr. med, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UiO_IMUTI
Record Dates: First submitted 2013-04-04; First posted 2013-05-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Acute Cystitis (Excl in Pregnancy)
MeSH Terms: interventions — Ibuprofen; Amdinocillin; Amdinocillin Pivoxil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Active Comparator): Tablet, over capsulated, 600mg three times a day for three days.
  Interventions: Drug: Ibuprofen
- Mecillinam (Active Comparator): Tablet, over capsulated, 200mg three times a day for three days.
  Interventions: Drug: Mecillinam

INTERVENTIONS:
Drug: Ibuprofen
  Other Names: Ibux
  Arms: Ibuprofen
Drug: Mecillinam
  Other Names: Selexid; Penomax
  Arms: Mecillinam

SUMMARY:
Although uncomplicated cystitis is considered to be a mild condition and mostly self limiting, most patients who see a doctor will be treated with antibiotics. Antibiotics are known to give a quick relief of symptoms and shorten the course of the condition by a few days. The aim of this study is to evaluate ibuprofen versus mecillinam in the treatment of uncomplicated cystitis in otherwise healthy, non-pregnant women. Our main objective is to see whether symptomatic treatment with ibuprofen is equally efficient as treatment with mecillinam in this group.

DETAILED DESCRIPTION:
The design of the study will be a double blinded randomized controlled trial (RCT). Half of the patients will receive treatment with mecillinam and the other half will receive treatment with ibuprofen. The study will follow the principles of Good Clinical Practice (GCP).

Urine cultures will be obtained on day one and after two weeks. The patients will be given a diary where they daily will register symptom load, possible complications or adverse effects and on which day they feel completely cured. We will contact the patients after two weeks to make sure they have followed the study procedures. After four weeks we will perform a final interview with the patient.

ELIGIBILITY:
Inclusion Criteria:

* woman between 18 and 60 years of age
* dysuria and pollakiuria and/or urinary urgency
* ability to give written consent

Exclusion Criteria:

* pregnancy/breastfeeding child under one month of age
* diabetes
* kidney disease
* organic aciduria
* clinical suspicion of pyelonephritis; fever, reduced general condition, upper back pain
* vaginal symptoms such as discharge or irritation
* severe abdominal pain
* symptoms that have lasted for more than seven days
* one or more urinary tract infections within the lasts four weeks
* permanent bladder catheter or use of bladder catheter within the last four weeks
* use of antibiotics within the last two weeks
* participated in a clinical trial within the last four weeks
* previously undergone a pyelonephritis
* previous allergic reaction to penicillin
* previous allergic reaction to ibuprofen, or worsening of asthma when using nonsteroidal antiinflammatory drugs(NSAIDs)
* narrow oesophagus
* use of the drug probenecid
* severe gastritis or previous ulcer
* anticoagulative treatment
* ongoing use of steroids
* use of immunosuppressant drugs
* thrombocytopenia,
* Chrohn's disease or Ulcerative colitis
* heart insufficiency
* severe psychiatric illness or dementia
* severe drug addiction
* unable to communicate in Norwegian, Swedish or Danish language

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 383 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who are symptom free by day four | Four days
  Both symptom load with regard to specific symptoms and when feeling completely symptom free will be registered in the patient diary.

SECONDARY OUTCOMES:
The patients' symptom load with regard to specific symptoms. | Seven days
  Specific symptoms, such as dysuria, urgency and pollakiuria, will be given a number from 0-6 in the patient diary, 0 = no problem and 6= as bad as it can get.

OTHER OUTCOMES:
Proportion of patients who were in need of a secondary medical consult within the study period. | 28 days
Proportion of patients who developed an upper urinary tract infection (pyelonephritis). | 14 days
Proportion of patients who experienced severe adverse effects. | Seven days
Proportion of patients who had a relapse of symptoms within four weeks after being included in the study. | 28 days
Proportion of patients with a positive urine culture after four weeks. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lindbæk, Professor, Principal Investigator — University of Oslo, faculty of medicine, institute for health and society, department of general medicine, antibiotic centre of primary care
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Sachdeva A, Rai BP, Veeratterapillay R, Harding C, Nambiar A. Non-steroidal anti-inflammatory drugs for treating symptomatic uncomplicated urinary tract infections in non-pregnant adult women. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD014762. doi: 10.1002/14651858.CD014762.pub2. PMID 39698942
- [Derived] Vik I, Mdala I, Bollestad M, Cordoba GC, Bjerrum L, Neumark T, Damsgaard E, Baerheim A, Grude N, Lindbaek M. Predicting the use of antibiotics after initial symptomatic treatment of an uncomplicated urinary tract infection: analyses performed after a randomised controlled trial. BMJ Open. 2020 Aug 30;10(8):e035074. doi: 10.1136/bmjopen-2019-035074. PMID 32868350
- [Derived] Vik I, Bollestad M, Grude N, Baerheim A, Damsgaard E, Neumark T, Bjerrum L, Cordoba G, Olsen IC, Lindbaek M. Ibuprofen versus pivmecillinam for uncomplicated urinary tract infection in women-A double-blind, randomized non-inferiority trial. PLoS Med. 2018 May 15;15(5):e1002569. doi: 10.1371/journal.pmed.1002569. eCollection 2018 May. PMID 29763434
- [Derived] Vik I, Bollestad M, Grude N, Baerheim A, Molstad S, Bjerrum L, Lindbaek M. Ibuprofen versus mecillinam for uncomplicated cystitis--a randomized controlled trial study protocol. BMC Infect Dis. 2014 Dec 17;14:693. doi: 10.1186/s12879-014-0693-y. PMID 25516016